CLINICAL TRIAL: NCT04264169
Title: Risk Factors for Occurrence of Placenta Accrete Spectrum Following Primary Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Taman, lecturer, Mansoura University Hospital
Other Study IDs: R.19.12.685
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Placenta Accreta
Keywords: placenta accrete spectrum; ultrasound; Risk factors
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week

GROUPS / COHORTS (2):
- • Study group: 100 patients' attending to the antenatal care clinic for elective termination of pregnancy with history of previous one cesarean delivery and the current pregnancy will be complicated by placenta accreta spectrum
- • Control group: 100 patients' attending to the antenatal care clinic for elective termination of pregnancy with history of previous one cesarean delivery and the current pregnancy will not be complicated by placenta accreta spectrum

SUMMARY:
This study will be conducted on a group of patients undergoing repeat elective caesarean delivery attending at Mansoura university hospital.

- This study will investigate patients' attending to the antenatal care clinic for elective termination of pregnancy with history of previous one caesarean delivery in the period between (January 2020 till January 2021).

DETAILED DESCRIPTION:
Participants in this study will be a group of patients with past history of previous one caesarean delivery and attending for elective termination of the current pregnancy.

Patients data will be collected and analysed as following:

* Personal data: Age, residency, job, special habits, BMI
* Past obstetric history:

Gravidity, parity, full term normal delivery, full term assisted vaginal deliveries, preterm, stillbirth, abortion, previous pregnancy complication and complication during puerperium • Previous delivery: Indication, duration, place of delivery, results of delivery, complication during labour, complication during puerperium

* Past medical, surgical or gynaecological history
* Pregnancy by assisted reproductive techniques
* Current pregnancy complications
* Trans abdominal and trans vaginal ultrasound examination Patients will be considered to have placenta praevia if the lower edge of the placenta is less than 2 cm form the internal os of the cervix

Placenta accreta will be considered as the following(7, 8) (Placental lacunae, Loss of hypoechoic space, Abnormalities of uterus-bladder interface, Color Doppler abnormalities)

2D grey-scale Loss of the "clear zone" Loss or irregularity of the hypoechoic plane in the myometrium underneath the placental bed (the "clear zone") Abnormal placental lacunae Presence of numerous lacunae including some that are large and irregular (Fin berg grade 3) often containing turbulent flow visible in grey-scale imaging Bladder wall interruption Loss or interruption of the bright bladder wall (the hyperechoic band or "line" between the uterine serosa and the bladder lumen) Myometrial thinning Thinning of the myometrium overlying the placenta to <1 mm or undetectable Placental bulge Deviation of the uterine serosa away from the expected plane, caused by an abnormal bulge of placental tissue into a neighbouring organ, typically the bladder. The uterine serosa appears intact but the outline shape is distorted Focal exophytic mass Placental tissue seen breaking through the uterine serosa and extending beyond it. Most often seen inside a filled urinary bladder Color Doppler imaging Uterovesical hypervascularity Striking amount of colour Doppler signal seen between the myometrium and the posterior wall of the bladder. This sign probably indicates numerous, closely packed, tortuous vessels in that region (demonstrating multi-directional flow and aliasing artifact) Subplacental hypervascularity Striking amount of color Doppler signal seen in the placental bed. This sign probably indicates numerous,closely packed, tortuous vessels in that region (demonstrating multidirectional flow and aliasing artifact)

Bridging vessels Vessels appearing to extend from the placenta across the myometrium and beyond the serosa into the bladder or other organs. Often running perpendicular to the myometrium

Placental lacunae feeder vessels Vessels with high velocity blood flow leading from the myometrium into the placental lacunae, causing turbulence upon entry

At laparotomy the following data will be reviewed(6):

Grade 1: Abnormally adherent placenta (placenta adherenta or accreta)

* Macroscopically, the uterus shows no obvious distension over the placental bed (placental "bulge"), no placental tissue is seen invading through the surface of the uterus, and there is no or minimal neovascularity Grade 2: Abnormally invasive placenta (Increta)
* Abnormal macroscopic findings over the placental bed: bluish/purple colouring, distension (placental "bulge")
* Significant amounts of hypervascularity (dense tangled bed of vessels or multiple vessels running parallel craniocaudially in the uterine serosa)
* No placental tissue seen to be invading through the uterine serosa.
* Gentle cord traction results in the uterus being pulled inwards without separation of the placenta (so-called the dimple sign) Histologic criteria

  * Hysterectomy specimen or partial myometrial resection of the increta area shows placental villi within the muscular fibers and sometimes in the lumen of the deep uterine vasculature (radial or arcuate arteries) Grade 3: Abnormally invasive placenta (Percreta) Grade 3a: Limited to the uterine serosa Clinical criteria
  * At laparotomy
* Abnormal macroscopic findings on uterine serosal surface (as above) and placental tissue seen to be invading through the surface of the uterus
* No invasion into any other organ, including the posterior wall of the bladder (a clear surgical plane can be identified between the bladder and uterus)

  • Histologic criteria
* Hysterectomy specimen showing villous tissue within or breaching the uterine serosa Grade 3b: With urinary bladder invasion Clinical criteria

  • At laparotomy
* Placental villi are seen to be invading into the bladder but no other organs
* Clear surgical plane cannot be identified between the bladder and uterus Histologic criteria

  * Hysterectomy specimen showing villous tissue breaching the uterine serosa and invading the bladder wall tissue or urothelium Grade 3c: With invasion of other pelvic tissue/organs Clinical criteria
  * At laparotomy
* Placental villi are seen to be invading into the broad ligament, vaginal wall, pelvic sidewall or any other pelvic organ (with or without invasion of the bladder) Histologic criteria • Hysterectomy specimen showing villous tissue breaching the uterine serosa and invading pelvic tissues/organs (with or without invasion of the bladder) .For the purposes of this classification, "uterus" includes the uterine body and uterine cervix .

  * The data will be analysed after putting it in the following groups,
  * study group consisted of patients with placenta praevia diagnosed by TVUS, control group consisted of patients undergoing elective caesarean delivery without having placenta praevia by transvaginal ultrasound (TVUS) examination

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of previous one caesarean delivery
* Patients who refused trail of vaginal birth after caesarean section
* Patients with permanent indication for caesarean section like contracted pelvis
* Patient without any history of medical diseases

Exclusion Criteria:

* Patients with history of more than one previous caesarean delivery
* Patients with medical disorders complicating pregnancy kike preeclampsia and gestational diabetes mellitus
* Patients with known uterine abnormalities eg (Bicornuate uterus, Adenomyosis, Submucous fibroids and Myotonic dystrophy)
* Patients who are candidates for vaginal birth after caesarean section

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be conducted on a group of patients undergoing repeat elective cesarean delivery attending at Mansoura university hospital.
  - This study will investigate patients' attending to the antenatal care clinic for elective termination of pregnancy with history of previous one cesarean delivery
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
association between indication of primary Cesarean delivery and degree of severity of placenta accreta spectrum | 1 day
  association between indication of primary Cesarean delivery and degree of severity of placenta accreta spectrum

SECONDARY OUTCOMES:
the association between parity, gravidity, place of the primary Cesarean delivery, assisted conception, and vaginal delivery before and after the primary Cesarean delivery,postpartum complications and degree of placenta accreta spectrum | 1 week
  the association between parity, gravidity, place of the primary Cesarean delivery, assisted conception, and vaginal delivery before and after the primary Cesarean delivery ,postpartum complications and degree of placenta accreta spectrum

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Taman, MD, Principal Investigator — Faculty of Medicine - Mansoura University
Locations (1):
- Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauniaux E, Chantraine F, Silver RM, Langhoff-Roos J; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Epidemiology. Int J Gynaecol Obstet. 2018 Mar;140(3):265-273. doi: 10.1002/ijgo.12407. No abstract available. PMID 29405321